CLINICAL TRIAL: NCT02627742
Title: Evaluation of a Practice Change to Include The MetaNeb® System to Reduce Postoperative Pulmonary Complications
Brief Title: Evaluation of The MetaNeb® System to Reduce Postoperative Pulmonary Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Organization: Baxter Healthcare Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR-RR2015-001
Record Dates: First submitted 2015-12-02; First posted 2015-12-11 (Estimated); Results first posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Atelectasis; Pulmonary Complications
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- METANEB (Experimental): Patients will receive standard care with the addition of therapy with The MetaNeb® System.
  Interventions: Device: MetaNeb® System

INTERVENTIONS:
Device: MetaNeb® System — The treatment protocol used for Respiratory Care during the CHANGE IN PRACTICE period of the Study will be that prescribed by the patient's health care team in the routine standard care of each patient. With the exception of standard airway clearance and lung expansion procedures, other components of the patients respiratory care regimen will remain the same as during the standard therapy period, however the CHANGE IN PRACTICE will incorporate the use/treatment with The MetaNeb® System as an alternative to usual airway clearance and lung expansion procedures. Use of The MetaNeb® System will follow the labeling of the device.

SUMMARY:
To determine if a therapy regimen including treatment with The MetaNeb® System had a positive impact on the rate of pulmonary complications related to atelectasis and/or secretion retention that occur in high risk post-operative patients. This is a non-randomized facility (or hospital) level pre-post intervention study.

DETAILED DESCRIPTION:
Post-operative pulmonary complications (PPC) are associated with significant excess morbidity, mortality and healthcare expenditure. Although PPCs are an incompletely understood multifactorial syndrome, atelectasis is recognized as a critical component. A variety of strategies have been shown to reduce the risk for development of post-operative atelectasis including lung expansion (LE) therapies. Well-designed studies are needed to distinguish which LE approach has the greatest potential to optimize patient care, clinical outcomes and cost savings.

Intrapulmonary percussive ventilation (IPV) devices have been in use for more than 25 years and are used widely in the acute care, post-surgical, and homecare setting. Such devices provide both LE and airway clearance therapy (ACT) for patients with obstructive and/or restrictive lung diseases and conditions. The MetaNeb® System is an LE expansion modality that incorporates all the physiological effects of IPV while providing additional therapeutic advantages intended primarily to more effectively treat or prevent pulmonary atelectasis.

The study was be conducted in two stages. In Stage I of the study, a retrospective review of medical records for post-surgical patients, who received STANDARD THERAPY as defined by current hospital and respiratory care department policies and procedures was performed. In Stage II, a CHANGE IN PRACTICE was made and patients received standard care with the addition of therapy with The MetaNeb® System. Demographic, clinical & outcome data was collected for eligible patients during the two stages of the study. Study staff collected data from the medical records, following a protocol determined schedule.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Post-thoracic, -upper abdominal or -aortic surgery Open surgical procedure Incision at or above the umbilicus

High risk defined by:

Documented ASA class ≥ 3 OR

Documented ASA class 2 AND One or more of the following:

Current smoker or smoking history within past 6 months History of COPD Documented obesity and/or BMI ≥ 30 kg/m2 Age ≥ 75

Exclusion Criteria:

Contraindication to Continuous High Frequency Oscillation (CHFO) therapy

Minimally invasive, or ". . . scopic" procedure.

Spinal surgery involving a posterior approach.

Surgery for organ transplant.

Chronic invasive positive pressure ventilation (PPV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Liesching, MD, FCCP, Principal Investigator — Lahey Hospital & Medical Center; Maurizio Cereda, MD, Principal Investigator — University of Pennsylvania; Toan Huynh, MD FACS FCCM, Principal Investigator — Carolinas Medical Center
Locations (3):
- United States (3):
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Carolinas Medical Center, Charlotte, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Huynh TT. et al.,
- [Derived] Huynh TT, Liesching TN, Cereda M, Lei Y, Frazer MJ, Nahouraii MR, Diette GB. Efficacy of Oscillation and Lung Expansion in Reducing Postoperative Pulmonary Complication. J Am Coll Surg. 2019 Nov;229(5):458-466.e1. doi: 10.1016/j.jamcollsurg.2019.06.004. Epub 2019 Jul 27. PMID 31362061

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Therapy - Stage I: Retrospectively collected medical records related to respiratory care from patients on STANDARD THERAPY without MetaNeb® as defined by current hospital and Respiratory Care department policies and procedures, was conducted. The purpose of Stage I was to estimate the incidence of postoperative pulmonary complications that occur in postsurgical patients who received standard therapy.
- Change in Practice - Stage II: Patients who received standard care with the addition of therapy with The MetaNeb® System.
  MetaNeb® System: The treatment protocol used for Respiratory Care during the CHANGE IN PRACTICE period of the Study was that prescribed by the patient's health care team in the routine standard care of each patient. With the exception of standard airway clearance and lung expansion procedures, other components of the patient's respiratory care regimen remained the same as during the standard therapy period, however the CHANGE IN PRACTICE incorporated the use/treatment with The MetaNeb® System as an alternative to usual airway clearance and lung expansion procedures. Use of The MetaNeb® System followed the labeling of the device.
Period: Overall Study
Arm/Group | Standard Therapy - Stage I | Change in Practice - Stage II
Started | 210 | 209
Completed | 201 | 202
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Therapy - Stage I | Change in Practice - Stage II | Total
Number analyzed (Participants) | 210 | 209 | 419
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 129 | 113 | 242
  >=65 years | 81 | 96 | 177
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.4 (15.48) | 61.1 (13.72) | 59.24 (14.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 78 | 173
  Male | 115 | 131 | 246
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 203 | 201 | 404
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 29 | 61
  White | 168 | 177 | 345
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Significant Postoperative Pulmonary Complication Incidence.
Description: One or more of the following that occurs within seven (7) days of the post-surgical admission will be considered a Significant Postoperative Pulmonary Complication (PPC)
  * Patient requires prolonged mechanical ventilation (> 24 hours from post-surgical admission)
  * Patient requires prolonged respiratory support for > 24 hours from post-surgical admission
  * Diagnosis of pneumonia within seven (7) days
  * Readmission to ICU for pulmonary complications within seven (7) days of post-surgical hospital admission
Time Frame: Within seven (7) days of the post-surgical admission
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Therapy - Stage I | Change in Practice - Stage II
Number analyzed (Participants) | 210 | 209
Participants
  Number of subjects with ≥ 1 PPC | 48 | 33
  Number of subjects without ≥ 1 PPC | 162 | 176

2. Secondary Outcome: Requirement for Invasive Mechanical Ventilation for > 48 Hours Within Seven (7) Days of the Post-surgical Hospital Admission
Description: Defined as patient requirement for invasive mechanical ventilation (MV) for > 48 hours (after hour 48) post-operatively. This includes patients that require re-intubation after hour 48, regardless of length of time on MV in the first 48 hours postoperatively.
Time Frame: 7 days (From the time of post-surgical admission to the hospital through day 7 following the initial post-surgical admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Therapy - Stage I | Change in Practice - Stage II
Number analyzed (Participants) | 210 | 209
Participants | 19 | 14

3. Secondary Outcome: Requirement for Respiratory Support > 48 Hours Within Seven (7) Days of the Post-surgical Hospital Admission
Description: Respiratory support greater than the patient's baseline level for a period longer than 48 hours
  * Requirement for non-invasive ventilation (NIV) above patient's baseline requirement after hour 48 from post-surgical admission or continuous positive airway pressure (CPAP) above patient's baseline requirement after hour 48.
  * Requirement for O2 therapy > 40 % FiO2 or > 5 LPM pm via Nasal Cannula (and above patient's baseline) after hour 48 postoperatively.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Therapy - Stage I | Change in Practice - Stage II
Number analyzed (Participants) | 210 | 209
Participants | 21 | 19

4. Secondary Outcome: Length of ICU Stay During Initial Hospital Stay
Description: ICU length of stay, during initial hospital stay, was determined by calculating the number of days/hours spent in ICU. The following was documented:
  * Time of admission to the ICU to actual time of initial discharge from the ICU during initial hospital stay
  * Total ICU days/hours (includes readmissions) during initial hospital stay
Time Frame: Total days/hours until time of discharge from the hospital, up to 8 weeks
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard Therapy - Stage I | Change in Practice - Stage II
Number analyzed (Participants) | 210 | 209
Days | 2.11 (6.004) | 1.27 (2.672)

5. Secondary Outcome: Length of Hospital Stay During Initial Hospital Stay
Description: Hospital length of stay was determined by calculating the number of days/hours spent in hospital. The following was documented:
  • Time of admission to time of discharge from the hospital (total days/hours)
Time Frame: Time of admission until time of discharge from the hospital, up to 8 weeks
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard Therapy - Stage I | Change in Practice - Stage II
Number analyzed (Participants) | 210 | 209
Days | 8.40 (7.895) | 6.78 (4.978)

6. Secondary Outcome: Readmission to ICU and Transfers to Elevated Level of Care for Pulmonary Complications During Initial Hospital Stay
Description: Readmissions to ICU and transfers to an elevated level of care, during the initial hospital stay, was documented for each event. The following was documented:
  * Number of readmission to ICU or elevated level of care events
  * Number of patients requiring readmission to the ICU or to an elevated level of care
Time Frame: during hospital stay, up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Therapy - Stage I | Change in Practice - Stage II
Number analyzed (Participants) | 210 | 209
Participants
  Number of readmissions: None | 205 | 204
  Number of readmissions: Once | 5 | 4
  Number of readmissions: More than Once | 0 | 1

7. Secondary Outcome: Readmission to Hospital
Description: Hospital records were reviewed at each site, 30 days after the last patient has been discharged from the hospital. Readmissions, for any cause, within 30 days of discharge for any study patient were documented.
Time Frame: 30 days following discharge from the hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Therapy - Stage I | Change in Practice - Stage II
Number analyzed (Participants) | 210 | 209
Participants | 36 | 28

8. Secondary Outcome: Time on Mechanical Ventilation
Description: * Time to initial extubation from time of initial intubation, if initial intubation was placed after surgery; or from time of post-surgical admission, if intubation was in place prior to start of surgery
  * Total time on invasive mechanical ventilation - was determined for each patient by calculating the total number of days/hours intubated and mechanically ventilated from the time of post-surgical admission until the time of initial hospital discharge.
  * Total time on non-invasive ventilation - was determined for each patient by calculating the total number of days/hours ordered for non-invasive ventilation from the time of post-surgical admission to the hospital unit until the time of initial hospital discharge.
Time Frame: total hours/days from the time of the post-surgical admission to the hospital unit until time of discharge from the hospital, up to 8 weeks
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Standard Therapy - Stage I | Change in Practice - Stage II
Number analyzed (Participants) | 210 | 209
Hours
  Time to Initial Extubation | 18.57 (75.04) | 7.64 (25.02)
  Total Time on Invasive Mechanical Ventilation | 23.7 (107.47) | 8.5 (27.40)
  Total Time on Non-Invasive Mechanical Ventilation | 0.5 (4.21) | 0.6 (3.31)

ADVERSE EVENTS:
Time Frame: Screening up to 8 weeks post-surgery
Arm/Group | Standard Therapy - Stage I | Change in Practice - Stage II
All-Cause Mortality (participants affected / at risk) | 9/210 | 7/209
Serious Adverse Events (participants affected / at risk) | 9/210 | 8/209
Other Adverse Events (participants affected / at risk) | 0/210 | 1/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Therapy - Stage I (N=210) | Change in Practice - Stage II (N=209)
Complications from pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intra-abdominal infection from untreated DLBCL (General disorders) | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Cardiomyopathy; cardiac arrest (Cardiac disorders) | 1 | 0
Inflammatory response syndrome due to aortic aneurysm (Vascular disorders) | 1 | 0
Cardiorespiratory failure (Cardiac disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemorrhage- intracranial NOS, hemorrhage (Nervous system disorders) | 1 | 0
Respiratory arrest, hepatic failure (General disorders) | 1 | 0
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diffuse anoxic brain injury (Nervous system disorders) | 0 | 1
Cardiac arrest, cause unspecified (Cardiac disorders) | 0 | 1
Cardiac death (General disorders) | 0 | 1
Cause of death is unknown (General disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Therapy - Stage I (N=210) | Change in Practice - Stage II (N=209)
Intolerant to device with agitation, increased work of breathing (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT02627742/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT02627742/SAP_001.pdf